CLINICAL TRIAL: NCT04379154
Title: Analysis of Volatile Organic Compounds by Electronic Noses in Hospitalised Patients for an Infection by (SARS-CoV-2): Predictive Interest in Short-term Evolution
Brief Title: Analysis of Volatile Organic Compounds by Electronic Noses in Hospitalised Patients for an Infection by SARS-COV-2 (COVID-19)
Acronym: VOC-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020_0060
Record Dates: First submitted 2020-04-28; First posted 2020-05-07 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Volatile Organic Compounds analysis (Experimental): Volatile Organic Compounds analysis in exhaled air in patients hospitalised for COVID-19 infection
  Interventions: Device: Volatile Organic Compounds analysis

INTERVENTIONS:
Device: Volatile Organic Compounds analysis — Volatile Organic Compounds analysis in exhaled air by electronic noses

SUMMARY:
The study of volatile organic compounds (VOCs) detected in exhaled air is an innovative research area for respiratory diseases. This analysis can be done by the technique of electronic nose, simpler and faster, which provides an idea of the general profile of the VOCs without identifying them. The VOCs in exhaled air in patients hospitalized for COVID-19 infection are analysed in this study, using electronic noses.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected by SARS-CoV-2 whose medical condition warrants hospitalisation (out of intensive care) for oxygen therapy less or equal to 4 l/min
* Patients must be 18 years of age or older
* Fluent in the French language
* Have signed a consent form
* Being affiliated with healthcare insurance

Exclusion Criteria:

* Pregnant woman
* Patient deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Profiles of volatile organic compounds (VOCs) in exhaled air between 2 health conditions | 1 day
  Comparison of variation of profiles of Volatile Organic Compounds in exhaled air from electronic noses (a set of sensors interacting with the VOCs exhaled). The analysis of the generated signal (resistance or load variations) is characteristic of the composition of VOCs), between patients who improve and patients who get worse during their hospitalisation for COVID-19 infection

SECONDARY OUTCOMES:
Profiles of volatile organic compounds (VOCs) in exhaled air on 1 health condition | 2 weeks
  Comparison of variation of profiles of Volatile Organic Compounds in exhaled air from electronic noses (a set of sensors interacting with the VOCs exhaled. The analysis of the generated signal (resistance or load variations) is characteristic of the composition of VOCs), between the start and the discharge to the hospital in patients infecting and recovering from COVID-19.
Profiles of volatile organic compounds (VOCs) in exhaled air between 2 periods | 4 months
  Comparison of variation of profiles of Volatile Organic Compounds in exhaled air from electronic noses (a set of sensors interacting with the VOCs exhaled. The analysis of the generated signal (resistance or load variations) is characteristic of the composition of VOCs), between the hospitalisation period and a post-hospitalisation follow-up consultation in patients infected by COVID-19 and recovered.
Profiles of volatile organic compounds (VOCs) in exhaled air by mass spectrometry at each visit based on patient evolution status. | 4 months
  Comparison of variation of profiles of Volatile Organic Compounds in exhaled air from mass spectrometry, at hospitalisation, post-hospitalisation and follow-up consultation in patients infected by COVID-19 and recovered.

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Salvator, Principal Investigator — Pneumology unit
Locations (1):
- Hôpital Foch, Suresnes, France